CLINICAL TRIAL: NCT05820412
Title: Individualized Use of a Multi-dimensional Instrumented Assessment of Motor Function and Balance Following an Intensive Therapy Episode of Care
Brief Title: Individualized Assessment of Motor Function and Balance in Intensive Therapy
Status: Completed | Type: Observational
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jamie Hall, Assistant Teaching Professor, University of Missouri-Columbia
Other Study IDs: 2096274
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neurodevelopmental Disorders
Keywords: technology; neurodevelopmental disorders; pediatrics; rehabilitation; intensive therapy
MeSH Terms: conditions — Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intensive interdisciplinary therapy — Intensive interdisciplinary therapy includes an intense burst of physical, occupational, and/or speech therapy with high intensity and frequency in a duration (e.g. 3-6 hours/day, 3-5 days/week for 4 weeks)

SUMMARY:
The goal of this study is to assess the individualized use of technology to assess motor function and balance for ambulatory children participating in an intensive therapy episode of care and determine the effectiveness of the program. Children 7-17 years old who can walk and are completing an intensive therapy episode of care will be recruited to participate in this study. Demographic, health history, and PT,OT,ST medical records will be collected. Based on the participant's functional goals, motor function and balance tests will be selected including common balance tests (standing with eyes open, standing with eyes closed), walking, walking and turning, standing up and sitting down from a bench, reaction time, and step down. Participants will be tested before, immediately after, 6 weeks after, and 12 weeks after the episode of care.

DETAILED DESCRIPTION:
The goal of this study is to assess the individualized use of instrumented assessment of motor function and balance for ambulatory children participating in an intensive therapy episode of care and determine the effectiveness of the intervention. Children 7-17 with neurodevelopmental diagnosis, GMFCS Levels I and II and completing an intensive therapy episode of care will be recruited to participate in this study. Demographic, health history, and PT,OT,ST medical records will be collected. Based on the participant's functional goals, motor function and balance tests in single and dual conditions will be selected including Romberg balance tests, walking, walking and turning, sit to/from stand, reaction time, and step down administered while participant is recorded using a portable measurement platform which incorporates a custom force plate, Azure Kinect spatial sensor, and interface board. Participants will be tested before, immediately after, 6 weeks after, and 12 weeks after the episode of care. Testing is estimated to last for 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory children 7-17 years old receiving care in an interdisciplinary, intensive therapy program
* GMFCS Levels I and II
* able to follow 2-3 step directions
* English speaking

Exclusion Criteria:

* orthopedic surgery in the past year or
* significant visual impairment
* significant hearing impairment.

Ages: 7 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: Ambulatory children aged 7-17 years old receiving care in an interdisciplinary intensive therapy program.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Eyes closed standing on firm surface | before physical therapy begins
  center of pressure as a measure of postural control obtained from a forceplate obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | immediately following physical therapy
  center of pressure as a measure of postural control obtained from a forceplate obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | 6 weeks following physical therapy
  center of pressure as a measure of postural control obtained from a forceplate obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | 12 weeks following physical therapy
  center of pressure as a measure of postural control obtained from a forceplate obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | before physical therapy
  joint kinematics (movement strategies) obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | immediately following physical therapy
  joint kinematics (movement strategies) obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | 6 weeks following physical therapy
  joint kinematics (movement strategies) obtained while eyes closed standing on firm surface
Eyes closed standing on firm surface | 12 weeks following physical therapy
  joint kinematics (movement strategies) obtained while eyes closed standing on firm surface
Walking | before physical therapy
  speed obtained from spatial sensor
Walking | immediately following physical therapy
  speed obtained from spatial sensor
Walking | 6 weeks following physical therapy
  speed obtained from spatial sensor
Walking | 12 weeks following
  speed obtained from spatial sensor
Walking | before physical therapy
  stride length obtained from spatial sensor
Walking | immediately following physical therapy
  stride length obtained from spatial sensor
Walking | 6 weeks following physical therapy
  stride length obtained from spatial sensor
Walking | 12 weeks following physical therapy
  stride length obtained from spatial sensor
5 Times sit to stand test | before physical therapy
  time to complete obtained from spatial sensor
5 Times sit to stand test | immediately following physical therapy
  time to complete obtained from spatial sensor
5 Times sit to stand test | 6 weeks following physical therapy
  time to complete obtained from spatial sensor
5 Times sit to stand test | 12 weeks following physical therapy
  time to complete obtained from spatial sensor
5 Times sit to stand test | before physical therapy
  knee joint kinematics obtained from spatial sensor
5 Times sit to stand test | immediately following physical therapy
  knee joint kinematics obtained from spatial sensor
5 Times sit to stand test | 6 weeks following physical therapy
  knee joint kinematics obtained from spatial sensor
5 Times sit to stand test | 12 weeks following physical therapy
  knee joint kinematics obtained from spatial sensor
Step down | before physical therapy
  knee joint kinematics obtained from spatial sensor
Step down | immediately following physical therapy
  knee joint kinematics obtained from spatial sensor
Step down | 6 weeks following physical therapy
  knee joint kinematics obtained from spatial sensor
Step down | 12 weeks following physical therapy
  knee joint kinematics obtained from spatial sensor

SECONDARY OUTCOMES:
Measures of processes of care | immediately following the episode of care
  Questionnaire designed to assess parents' perceptions of the care they and their children receive from children's rehabilitation treatment centres. It is a means to assess family-centred behaviours of health care providers.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Therapy Center--MU Healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hall JB, Chole D, Pruitt TC, Linkeman K. Caregiver Perceptions of an Interdisciplinary Intensive Therapy Program: A Qualitative Study. Pediatr Phys Ther. 2023 Apr 1;35(2):228-235. doi: 10.1097/PEP.0000000000000994. Epub 2023 Jan 10. PMID 36637445
- [Background] Guess TM, Bliss R, Hall JB, Kiselica AM. Comparison of Azure Kinect overground gait spatiotemporal parameters to marker based optical motion capture. Gait Posture. 2022 Jul;96:130-136. doi: 10.1016/j.gaitpost.2022.05.021. Epub 2022 May 21. PMID 35635988
- [Background] Thomas J, Hall JB, Bliss R, Guess TM. Comparison of Azure Kinect and optical retroreflective motion capture for kinematic and spatiotemporal evaluation of the sit-to-stand test. Gait Posture. 2022 May;94:153-159. doi: 10.1016/j.gaitpost.2022.03.011. Epub 2022 Mar 21. PMID 35334335
- [Background] French MA, Roemmich RT, Daley K, Beier M, Penttinen S, Raghavan P, Searson P, Wegener S, Celnik P. Precision Rehabilitation: Optimizing Function, Adding Value to Health Care. Arch Phys Med Rehabil. 2022 Jun;103(6):1233-1239. doi: 10.1016/j.apmr.2022.01.154. Epub 2022 Feb 15. PMID 35181267
- [Background] Gannotti ME. Coupling Timing of Interventions With Dose to Optimize Plasticity and Participation in Pediatric Neurologic Populations. Pediatr Phys Ther. 2017 Jul;29 Suppl 3(Suppl 3 IV STEP 2016 CONFERENCE PROCEEDINGS ):S37-S47. doi: 10.1097/PEP.0000000000000383. PMID 28654476
- [Background] Gannotti ME, Christy JB, Heathcock JC, Kolobe TH. A path model for evaluating dosing parameters for children with cerebral palsy. Phys Ther. 2014 Mar;94(3):411-21. doi: 10.2522/ptj.20130022. Epub 2013 Nov 14. PMID 24231231
- [Background] Tinderholt Myrhaug H, Ostensjo S, Larun L, Odgaard-Jensen J, Jahnsen R. Intensive training of motor function and functional skills among young children with cerebral palsy: a systematic review and meta-analysis. BMC Pediatr. 2014 Dec 5;14:292. doi: 10.1186/s12887-014-0292-5. PMID 25475608